CLINICAL TRIAL: NCT03769922
Title: The MESOCOLIC Trial: Mesenteric Excision Surgery or Conservative Limited Resection in Crohn's Disease
Brief Title: Postoperative Progression of the Disease Following Extensive Versus Limited Mesenteric Excision for Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: University Hospital of Limerick (Other); The Cleveland Clinic (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Weiming Zhu, Chief of general surgery, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018NZKY-025-02
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Surgical Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extensive mesenteric resection (Experimental): Mesenteric is resected avoiding the root region, i.e. 1 cm from the root of ileocolic artery and vein.
  Interventions: Procedure: Extensive mesenteric resection
- Limited mesenteric excision (Active Comparator): Mesentery is retained, i.e. "Close shave" or 3 cm from the border of bowel (using whatever approach - clips, or haemostatic vessel sealing device).
  Interventions: Procedure: Limited mesenteric excision

INTERVENTIONS:
Procedure: Extensive mesenteric resection — The mesentery is resected avoiding the root region.
  Arms: Extensive mesenteric resection
Procedure: Limited mesenteric excision — The mesentery is retained.
  Arms: Limited mesenteric excision

SUMMARY:
The study evaluates whether there is a reduction in the rate of postoperative progression of the disease following extensive mesenteric excision (EME), when compared to that of limited mesenteric excision (LME), in patients undergoing ileocolic resection for Crohn's disease. Half of participants will receive EME, while the other half will receive LME.

DETAILED DESCRIPTION:
EME and LME are the two surgical procedures which are commonly used in the treatment of Crohn's disease. However, the areas of the mesenteric tissue resected are different.

EME means that the mesentery is resected avoiding the root region, i.e. 1 cm from the root of ileocolic artery and vein.

LME represents that the mesentery is retained, i.e. "Close shave" or 3 cm from the border of bowel (using whatever approach - clips, or haemostatic vessel sealing device).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease limited to the distal ileum and/or right colon receiving their index ileocolonic resection
* Patients with a documented history of Crohn's disease based on endoscopic, radiological, or histological criteria

Exclusion Criteria:

* Pregnancy or willingness to become pregnant in the following year
* Previous ileocolic resection history
* Patients having Crohn's disease lesion at a gastrointestinal site other than the terminal ileum cecum, or right colon
* Patients having an internal fistula which required resection of another segment of bowel

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Accumulated 5-year postoperative surgical recurrence | 5 years after the first surgery
  The requirement for repeat surgery for a Crohn's disease related indication.

SECONDARY OUTCOMES:
Accumulated 5-year endoscopic recurrence | 5 years after the first surgery
  Disease proximal to the anastomosis or in the perianastomotic are considered to be a endoscopic recurrence (Rutgeert's score i2, or higher, disease in other sites is not considered recurrence)
Accumulated 5-year clinical recurrence | 5 years after the first surgery
  The presence of endoscopic disease (i2, or higher) or radiological evidence plus the presence of symptoms attributable to Crohn's disease that are severe enough to require medical or surgical treatment.

OTHER OUTCOMES:
postoperative operation-related complications | 30 day
  30-day postoperative morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Weiming, Principal Investigator — Jinling Hospital, Nanjing, China.; John Calvin Coffey, Principal Investigator — University Hospital Limerick, Limerick, Ireland.; Luca Stocchi, Principal Investigator — The Cleveland Clinic
Locations (1):
- General Hospital of Eastern Theater Command, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coffey CJ, Kiernan MG, Sahebally SM, Jarrar A, Burke JP, Kiely PA, Shen B, Waldron D, Peirce C, Moloney M, Skelly M, Tibbitts P, Hidayat H, Faul PN, Healy V, O'Leary PD, Walsh LG, Dockery P, O'Connell RP, Martin ST, Shanahan F, Fiocchi C, Dunne CP. Inclusion of the Mesentery in Ileocolic Resection for Crohn's Disease is Associated With Reduced Surgical Recurrence. J Crohns Colitis. 2018 Nov 9;12(10):1139-1150. doi: 10.1093/ecco-jcc/jjx187. PMID 29309546
- [Background] Li Y, Zhu W, Gong J, Zhang W, Gu L, Guo Z, Cao L, Shen B, Li N, Li J. Visceral fat area is associated with a high risk for early postoperative recurrence in Crohn's disease. Colorectal Dis. 2015 Mar;17(3):225-34. doi: 10.1111/codi.12798. PMID 25307174
- [Background] Li Y, Ge Y, Gong J, Zhu W, Cao L, Guo Z, Gu L, Li J. Mesenteric Lymphatic Vessel Density Is Associated with Disease Behavior and Postoperative Recurrence in Crohn's Disease. J Gastrointest Surg. 2018 Dec;22(12):2125-2132. doi: 10.1007/s11605-018-3884-9. Epub 2018 Jul 24. PMID 30043133
- [Derived] Li Y, Mohan H, Lan N, Wu X, Zhou W, Gong J, Shen B, Stocchi L, Coffey JC, Zhu W. Mesenteric excision surgery or conservative limited resection in Crohn's disease: study protocol for an international, multicenter, randomized controlled trial. Trials. 2020 Feb 21;21(1):210. doi: 10.1186/s13063-020-4105-x. PMID 32085793